CLINICAL TRIAL: NCT07090135
Title: Enhance the Restorative Power of Sleep Through TES-TI Power Naps
Brief Title: Power Nap With TES-TI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Corundum Convergence Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2025-0481; A538900 (Other: UW Madison); SMPH/PSYCHIATRY/PSYCHIATRY (Other: UW Madison); Protocol Version 12/18/25 (Other: UW Madison)
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Non-restorative Sleep; Healthy Volunteer
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Stimulation followed by no stimulation (Experimental): Participants will receive stimulation during their nap at the first visit, and no stimulation during their nap at the second visit.
  Interventions: Device: Transcranial electrical stimulation with Temporal Interference (TES-TI)
- No stimulation followed by stimulation (Experimental): Participants will not receive stimulation during their nap at the first visit, and receive stimulation during their nap at the second visit.
  Interventions: Device: Transcranial electrical stimulation with Temporal Interference (TES-TI)

INTERVENTIONS:
Device: Transcranial electrical stimulation with Temporal Interference (TES-TI) — TES-TI uses specific electrode arrangement patterns to selectively stimulate the brain. Participants will wear an hdEEG (high density electroencephalography) cap which will allow intermittent periods of stimulation from TES-TI.

SUMMARY:
The goal of this clinical trial is to find out whether stimulating the brain with electrical current during naps can increase certain kinds of brain activity that happen during sleep and lead to improvements in mental fatigue.

Participants will attend 2 study visits, each of which may last up to 4-5 hours. During these visits, participants will wear a high density electroencephalography (hdEEG) cap and take a nap.

DETAILED DESCRIPTION:
This project aims to use transcranial electrical stimulation with temporal interference (TES-TI) to enhance the production of sleep slow waves, boosting the restorative power of sleep and mitigating cognitive impairment (mental fatigue) and its underlying cause (brain fatigue).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-75 of any gender identity
* Self-reported non-restorative sleep, as measured by a REST-Q score
* English-speaking (able to provide consent and complete questionnaires)
* Capable of taking daytime naps
* US Citizen

Exclusion Criteria:

* Any current or history of neurological disorders or acquired neurological disease (e.g. stroke, traumatic brain injury), including intracranial lesions
* History of inpatient psychiatric hospitalization
* History of head trauma resulting in prolonged loss of consciousness; or a history of >3 grade I concussions
* Current history of poorly controlled headaches including intractable or poorly controlled migraines

  • Any systemic illness or unstable medical condition that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.)
* History of seizures, diagnosis of epilepsy, history of abnormal (epileptiform) EEG, or family history of treatment resistant epilepsy except for a single seizure of benign etiology (e.g. febrile seizures) in the judgment of a board-certified neurologist
* Possible pregnancy or plan to become pregnant in the next 6 months
* Any metal in the head
* Any medical devices or implants (i.e. cardiac pacemaker, medication infusion pump, cochlear implant, vagal nerve stimulator)
* Dental implants
* Permanent retainers
* Any hair braid, dreadlocks, hair pieces, or extensions which cannot be taken out before the study sessions
* Any head coverings or headdress that participant feels uncomfortable removing for the purposes of study sessions
* Any medication that may alter seizure threshold taken during the study i.e., ADHD stimulants (Adderall, amphetamine); Tricyclic/atypical antidepressants (amitriptyline, doxepine, imipramine, maprotiline, nortriptyline, bupropion); Antipsychotics (chlorpromazine, clozapine), Bronchodilators (theophylline, aminophylline); Antibiotics (fluoroquinolones, imipenem, penicillin, cephalosporins, metronidazole, isoniazid); Antivirals (valacyclovir, ritonavir); OTC antihistamines (diphenhydramine, Benadryl)
* Claustrophobia (a fear of small or closed places)
* Back problems that would prevent lying flat for up to two hours
* Regular night-shift work (second or third shift)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change in slow waves | Baseline to 1 month
  Researchers will do a power analysis on high density EEG data for slow wave frequency (3-5Hz) and see if there is increase in this frequency range during/post stimulation.
Change in sleep quality and mood | Baseline to 1 month
  Sleep quality and mood will be assessed using the Restorative Sleep Questionnaire (REST-Q), a 9-item questionnaire assessing aspects of restorative sleep. Each item is scored on a 5-point Likert scale, scores range from 9-45. A higher score indicates a more restorative sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Guilio Tononi, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes